CLINICAL TRIAL: NCT02255786
Title: Taking ACTion: Acceptance and Commitment Therapy for Parents of Children With Autism Spectrum Disorder
Brief Title: "ACT" for Parents of Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Organization for Autism Research (Other)
Responsible Party: Principal Investigator, Lisa A. Nowinski, PhD, Director, Neuropsychology Training, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P001563
Record Dates: First submitted 2014-09-15; First posted 2014-10-03 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Stress
Keywords: Group Therapy; Parents; Autism; Quality of Life
MeSH Terms: conditions — Autistic Disorder | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT Parent Group (Experimental): Participants will complete a total of five Acceptance and Commitment Therapy - Parent Group Sessions First four are held weekly, last session held one month from 4th session.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Treatment as Usual (No Intervention): Treatment as usual-Control

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and Commitment Therapy (ACT) is an intervention that fosters acceptance of uncomfortable thoughts and emotions as a coping strategy, and encourages engagement in valued behavior in the presence of these emotions. ACT has been successfully applied to parents of children with a variety of mental health presentations.
  Other Names: ACT
  Arms: ACT Parent Group

SUMMARY:
The investigators will develop and pilot test an intervention called "ACT for Parents" which aims to decrease stress and improve quality of life in parents of children < 15 years who have a diagnosis of autism spectrum disorder. A small randomized trial testing phase will be conducted to gather initial data on the treatment feasibility and acceptability, detect treatment effects between groups (ACT for Parents versus Treatment as Usual), and to refine the treatment design for a future clinical trial.

DETAILED DESCRIPTION:
Acceptance and Commitment Therapy (ACT) is an intervention that fosters acceptance of uncomfortable thoughts and emotions as a coping strategy, and encourages engagement in valued behavior in the presence of these emotions. ACT has been successfully applied to parents with similar mental health presentations. Using a randomized controlled study design, investigators seek to gather initial data on the treatment feasibility and acceptability, detect treatment effects in a cohort of parents who have a child (under the age of 15) with autism spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* A parent with a child (under the age of 15) with a diagnosis of Pervasive Developmental Disorder-NOS, Asperger's Disorder or Autistic Disorder
* Child with ASD diagnosed by a mental health or medical professional
* Must be comfortable speaking and reading and understanding English

Exclusion Criteria:

* Inability to attend sessions in person on the specified date/time/location of the intervention sessions
* unwillingness to be audio-taped should randomization into the experimental (ACT) group occur.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Acceptance and Action Questionnaire-II Score | From Basline to Month 2 (post-intervention) and from Month 2 to Month 3 (maintenance)
  The Acceptance and Action Questionnaire (AAQ-II, Bond et al., 2011) is a 10-item Likert scale that measures experiential acceptance (i.e., tendency to accept, rather than avoid, uncomfortable internal experiences) in adult samples.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Nowinski, PhD, Principal Investigator — Massachusetts General Hospital - Lurie Center; Kirstin Brown Birtwell, PhD, Study Director — Massachusetts General Hospital - Lurie Center
Locations (1):
- Lurie Center | Massachusetts General Hospital, Lexington, Massachusetts, United States